CLINICAL TRIAL: NCT00995618
Title: A Randomized, Double-Blind, Crossover, Pharmacodynamic and Pharmacokinetic Drug Interaction Study of Tranilast in Combination With Febuxostat Compared With Tranilast Alone and Febuxostat Alone in Healthy Subjects With Hyperuricemia
Brief Title: Study of Tranilast Alone or in Combination With Febuxostat in Patients With Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuon Therapeutics, Inc. (Industry)
Responsible Party: Nuon Therapeutics Clinical Trials Contact, Nuon Therapeutics
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A3006GT
Record Dates: First submitted 2009-10-06; First posted 2009-10-15 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Gout; Hyperuricemia
Keywords: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — tranilast; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranilast (Experimental): Tranilast tablets
  Interventions: Drug: Tranilast
- Febuxostat (Active Comparator): Febuxostat tablets
  Interventions: Drug: Febuxostat
- Combination (Experimental): Tranilast plus febuxostat
  Interventions: Drug: Combination - Tranilast and Febuxostat

INTERVENTIONS:
Drug: Tranilast — Tranilast tablets, 300 mg, QD
  Arms: Tranilast
Drug: Febuxostat — Febuxostat Tablets, 40 mg, QD
  Other Names: Uloric
  Arms: Febuxostat
Drug: Combination - Tranilast and Febuxostat — Tranilast, 300 mg QD; Febuxostat, 40 mg QD
  Arms: Combination

SUMMARY:
This is a randomized, double-blind, 3-period crossover phase 2 study in patients with documented hyperuricemia to evaluate the effect of tranilast on febuxostat pharmacokinetics (PK) and pharmacodynamics (PD) and to evaluate the effect of febuxostat on tranilast PK and PD as measured by reduction in serum uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 70
* Subjects with hyperuricemia who are otherwise healthy

Exclusion Criteria:

* Pregnant or nursing
* Known history of gout
* Clinically significant infection at Screening
* Known sensitivity to tranilast or febuxostat

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean decrease in serum uric acid levels | Seven days

SECONDARY OUTCOMES:
Analysis of pharmacokinetic parameters (AUC, Cmax) of tranilast, febuxostat and combination | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Director, Nuon Clinical Trials Group, Study Director — Nuon Therapeutics, Inc.
Locations (3):
- United States (3):
  - Nuon Investigative Site, Honolulu, Hawaii
  - Nuon Investigative Site, Evansville, Indiana
  - Nuon Investigative Site, Dallas, Texas